CLINICAL TRIAL: NCT01345175
Title: Randomized Control Trial Comparing Rifaximin and Placebo in the Treatment of Bowel Dysfunction After Anterior Resection for Rectal Cancer
Brief Title: Rifaximin and Placebo in the Treatment of Bowel Dysfunction After Anterior Resection for Rectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-045
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2023-03

CONDITIONS: Rectal Cancer
Keywords: rectal; colon; PLACEBO; RIFAXIMIN; metronidazole; 11-045
MeSH Terms: conditions — Rectal Neoplasms | interventions — Rifaximin; Metronidazole; Defecation; Prescriptions; Clinical Trials, Phase III as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pts receiving Rifaximin (Experimental): This group will receive rifaximin 400mg bid for 4 weeks. At 1 - 24 months after completion of the phase III portion of the trial, patients will be contacted by phone and given the option of receiving metronidazole in a followup, single arm study in which all patients receive the antibiotic. Patients who wish to participate will be mailed a drug prescription for a 3 week course of metronidazole 500mgs tid as well as the BFI forms and stool diary. Pretreatment and post treatment BFI scores will be collected and analyzed for change in bowel function as was done in the initial Phase III study.
  Interventions: Drug: Rifaximin
- Pts receiving placebo (Placebo Comparator): This group will receive a placebo bid for 4 weeks. At 1 - 24 months after completion of the phase III portion of the trial, patients will be contacted by phone and given the option of receiving metronidazole in a followup, single arm study in which all patients receive the antibiotic. Patients who wish to participate will be mailed a drug prescription for a 3 week course of metronidazole 500mgs tid as well as the BFI forms and stool diary. Pretreatment and post treatment BFI scores will be collected and analyzed for change in bowel function as was done in the initial Phase III study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — Pt will receive rifaximin 400mg bid for 4 weeks. Patients will at this stage on a volunteer basis be asked to submit stool samples and undertake a breath test. Patients will receive the respective treatment for four weeks. Following cessation of treatment all patients will be assessed using the BFI and respective patients will have repeat stool sampling and breath testing. Patients will then have these tests repeated 4 weeks later. This corresponds to 8 weeks after the start of the trial. For those patients not undertaking stool and breath testing, they will be reminded by phone, mail or email to fill out the BFI. Before and during the trial patients will be asked to fill out a weekly stool diary to evaluate trends on bowel function.
  Other Names: At 1 - 24 months after completion of the phase III portion of the trial, patients will be contacted by phone and given the option of receiving; metronidazole in a followup, single arm study in which all patients receive the antibiotic.; Patients who wish to participate will be mailed a drug prescription for a 3 week course of; metronidazole 500mgs tid as well as the BFI forms and stool diary. Pretreatment and; posttreatment BFI scores will be collected and analyzed for change in bowel function as; was done in the initial Phase III study.
  Arms: Pts receiving Rifaximin
Drug: Placebo — Pt will receive placebo bid for 4 weeks. Patients will at this stage on a volunteer basis be asked to submit stool samples and undertake a breath test. Patients will receive the respective treatment for four weeks. Following cessation of treatment all patients will be assessed using the BFI and respective patients will have repeat stool sampling and breath testing. Patients will then have these tests repeated 4 weeks later. This corresponds to 8 weeks after the start of the trial. For those patients not undertaking stool and breath testing, they will be reminded by phone, mail or email to fill out the BFI. Before and during the trial patients will be asked to fill out a weekly stool diary to evaluate trends on bowel function.
  Other Names: At 1 - 24 months after completion of the phase III portion of the trial,; patients will be contacted by phone and given the option of receiving; metronidazole in a followup, single arm study in which all patients receive; the antibiotic. Patients who wish to participate will be mailed a drug; prescription for a 3 week course of metronidazole 500mgs tid as well as the; BFI forms and stool diary. Pretreatment and post treatment BFI scores will be; collected and analyzed for change in bowel function as was done in the initial; Phase III study.
  Arms: Pts receiving placebo

SUMMARY:
The most common long-term problems after rectal surgery are bowel problems. These problems can include needing to pass bowel movements a lot, loose or mushy stools, inability to fully clear your bowels, and/or poor control of gas and stool. The investigators believe that a major cause of these problems is too much bacteria in the bowel and treatment with antibiotic tablets will hopefully help improve these bowel problems. In order to test this idea, the Colorectal Surgery Service of Memorial Sloan Kettering Cancer Center is sponsoring a clinical trial. This trial will compare the antibiotic rifaximin and a placebo (a harmless tablet that has no effect) in the treatment of these bowel problems. Following this we will attempt to see if another antibiotic metronidazole also helps to treat these bowel problems. Both Metronidazole and rifaximin are well established drugs that have minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of rectal cancer treated with an anterior resection preformed at MSKCC (tumor at or below 12cm from anal verge) with restoration of bowel continuity ≥1 and ≤ 5 years. (Patients may also have had procedures to construct neo-rectums including j-pouch, coloplasty, and end to side anastomosis).
* Patients ≥ 21 years of age.
* Presence of anterior resection symptoms by patients own assessment. These symptoms may include any of the following: incomplete evacuation, clustering of bowel motions, frequency of bowel motions, unformed stool, excessive flatus, or incontinence of flatus and/or feces.

Exclusion Criteria:

* Local recurrence of rectal cancer.
* Antibiotic treatment within the last 4 weeks for any condition.
* Pregnancy or breast feeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-04-26 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Paty, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pts Receiving Rifaximin | Pts Receiving Placebo
Started | 36 | 33
Completed | 30 | 27
Not Completed | 6 | 6
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Failed to complete BFI | 3 | 2
Not completed — Stopped taking medication | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pts Receiving Rifaximin | Pts Receiving Placebo | Total
Number analyzed (Participants) | 36 | 33 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.47 (8.87) | 61.09 (10.51) | 58.16 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 19 | 13 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 32 | 30 | 62
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 33 | 31 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 33 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed MSKCC Bowel Function Instrument (BFI Score) in Patients Following Anterior Resection (AR) or Sphincter Preserving Surgery (SPS) for Rectal Cancer.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pts Receiving Rifaximin | Pts Receiving Placebo
Number analyzed (Participants) | 36 | 33
Participants
  Completed BFI | 30 | 27
  Did not complete BFI | 6 | 6

2. Secondary Outcome: To Determine if Reduction in Intestinal Bacterial Quantity Correlates With Improvement in Bowel Symptoms (BFI Score).
Time Frame: 1 year
Population: N/A Data were not collected
Arm/Group | Pts Receiving Rifaximin | Pts Receiving Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: To Explore the Bacterial Composition of Stool Before and After Antibiotic Treatment.
Time Frame: 1 year
Population: N/A Data were not collected
Arm/Group | Pts Receiving Rifaximin | Pts Receiving Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Identify Dynamic Changes in Bowel Function During and After Antibiotic Treatment Using a Bowel Function Log.
Time Frame: 1 year
Population: N/A data were not completed
Arm/Group | Pts Receiving Rifaximin | Pts Receiving Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Efficacy of Metronidazole
Description: in the treatment of bowel dysfunction as measured by the MSKCC BFI in patients following AR or SPS for rectal cancer for patients who have no improvement following treatment with rifaximin or placebo.
Time Frame: 1 year
Population: N/A Data were not collected
Arm/Group | Pts Receiving Rifaximin | Pts Receiving Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Arm 1: Experimental: Pts Receiving Rifaximin: This group will receive rifaximin 400mg bid for 4 weeks. At 1 - 24 months after completion of the phase III portion of the trial, patients will be contacted by phone and given the option of receiving metronidazole in a followup, single arm study in which all patients receive the antibiotic. Patients who wish to participate will be mailed a drug prescription for a 3 week course of metronidazole 500mgs tid as well as the BFI forms and stool diary. Pretreatment and post treatment BFI scores will be collected and analyzed for change in bowel function as was done in the initial Phase III study.
  Rifaximin: Pt will receive rifaximin 400mg bid for 4 weeks. Patients will at this stage on a volunteer basis be asked to submit stool samples and undertake a breath test. Patients will receive the respective treatment for four weeks. Following cessation of treatment all patients will be assessed using the BFI and respective patients will have repeat stool sampling and breath testing. Patients will then have these tests repeated 4 weeks later. This corresponds to 8 weeks after the start of the trial. For those patients not undertaking stool and breath testing, they will be reminded by phone, mail or email to fill out the BFI. Before and during the trial patients will be asked to fill out a weekly stool diary to evaluate trends on bowel function.
- Arm 2: Placebo Comparator: Pts Receiving Placebo: This group will receive a placebo bid for 4 weeks. At 1 - 24 months after completion of the phase III portion of the trial, patients will be contacted by phone and given the option of receiving metronidazole in a followup, single arm study in which all patients receive the antibiotic. Patients who wish to participate will be mailed a drug prescription for a 3 week course of metronidazole 500mgs tid as well as the BFI forms and stool diary. Pretreatment and post treatment BFI scores will be collected and analyzed for change in bowel function as was done in the initial Phase III study.
  Placebo: Pt will receive placebo bid for 4 weeks. Patients will at this stage on a volunteer basis be asked to submit stool samples and undertake a breath test. Patients will receive the respective treatment for four weeks. Following cessation of treatment all patients will be assessed using the BFI and respective patients will have repeat stool sampling and breath testing. Patients will then have these tests repeated 4 weeks later. This corresponds to 8 weeks after the start of the trial. For those patients not undertaking stool and breath testing, they will be reminded by phone, mail or email to fill out the BFI. Before and during the trial patients will be asked to fill out a weekly stool diary to evaluate trends on bowel function.
Arm/Group | Arm 1: Experimental: Pts Receiving Rifaximin | Arm 2: Placebo Comparator: Pts Receiving Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/33
Other Adverse Events (participants affected / at risk) | 0/36 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Experimental: Pts Receiving Rifaximin (N=36) | Arm 2: Placebo Comparator: Pts Receiving Placebo (N=33)
Diarrhea (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT01345175/Prot_SAP_000.pdf